CLINICAL TRIAL: NCT05761899
Title: A First-In-Human Clinical Trial of Lentiviral-mediated CSF2RA Gene Transfer/Pulmonary Macrophage Transplantation Therapy of Hereditary Pulmonary Alveolar Proteinosis
Brief Title: Safety and Efficacy of PMT Therapy of hPAP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0424; R33HL156888 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Pulmonary Alveolar Proteinosis
Keywords: Pulmonary Alveolar Proteinosis; Pulmonary Macrophage Transplantation
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Gene-Corrected Macrophages (Experimental): Autologous bone marrow CD34+ cell-derived, CSF2RA lentiviral vector-transduced macrophages (CSF2RA gene-corrected macrophages) by bronchoscopic instillation into individual lung segments.
  Interventions: Combination Product: Gene-Corrected Macrophages administered by bronchoscopic instillation

INTERVENTIONS:
Combination Product: Gene-Corrected Macrophages administered by bronchoscopic instillation — This study will evaluate administration of autologous bone marrow CD34+ cell-derived, CSF2RA lentiviral vector-transduced macrophages (CSF2RA gene-corrected macrophages) by bronchoscopic instillation into individual lung segments on three occasions at 2-month intervals in patients with hPAP. The target (maximum) number of cells to be administered is 778 million gene-corrected macrophages per 70 kg patient, which is equal to 11.1 million cells/kg of ideal body weight.

SUMMARY:
The major goal of this study is to evaluate a new type of cell transplantation therapy for individuals with hereditary PAP, study a new treatment that may be useful for treatment of other diseases, and research mechanisms that drive the development and function of lung macrophages.

DETAILED DESCRIPTION:
Hereditary pulmonary alveolar proteinosis (hPAP) is a rare lung disease characterized by the progressive accumulation of pulmonary surfactant in alveoli resulting in progressive hypoxemic respiratory failure, and in some patients, secondary infections and/or pulmonary fibrosis. While hPAP affects men, women, and children, most patients present as children. The lung structure appears well-preserved in many cases with pathogenesis being driven by the consequences of the filling of alveoli with surfactant sediment; however, some patients develop respiratory failure caused by pulmonary fibrosis requiring therapeutic lung transplantation.

Hereditary PAP is caused by homozygous or compound heterozygous mutations in the genes (CSF2RA or CSF2RB) encoding the GM-CSF receptor alpha or beta chains, respectively. Mutations in these genes disrupt GM-CSF receptor function, blocking GM-CSF signaling and impairing the removal of excess surfactant from alveoli by alveolar macrophages (AMs).

This study is an open-label, non-randomized, single center clinical treatment study to evaluate the feasibility of manufacturing CSF2RA gene-corrected macrophages, as well as the safety, tolerability, efficacy, and durability of CSF2RA gene correction/pulmonary macrophage transplantation (PMT) therapy in three patients with hPAP caused by recessive homozygous or compound heterozygous CSF2RA mutations. In addition to safety and tolerability, the clinical trial will evaluate outcome measures related to clinical efficacy and biologic signature of CSF2RA gene-correction/PMT therapy, as well as pharmacokinetics, pharmacodynamics, and the mechanism of action.

The clinical trial design includes a 2-month observation period, a Baseline visit, 5-month treatment period, and Short-, Medium-, and Long-Term follow-up periods of 1, 4, and 10 years, respectively. Each patient will serve as their own self-control and receive a split-dose comprising three administrations of autologous, bone marrow cluster of differentiation 34+ (CD34+) cell-derived, lentiviral CSF2RA gene-corrected macrophages at a minimum of 2-month intervals, delivered by direct bronchoscopic instillation of cells into individual lung segments (5.8x105 cells/segment); an increasing number of cells at each administration will be achieved by sequentially increasing the number of segments treated. Current standard medical care (whole lung lavage and supplemental oxygen) will be continuously available to all enrolled patients.

Assessments will include safety (adverse events and serious adverse events), tolerability (short-term, treatment-emergent pulmonary symptoms), efficacy (beneficial effects on clinical, physiological, and radiological manifestations of hPAP), durability (persistence of beneficial effects), and mechanism of action (persistence, CSF2RA-expression, and function of alveolar macrophages (AMs)).

Expected results will inform the feasibility, safety, tolerability, efficacy, durability, and mechanism of action of gene transfer/PMT as therapy of hPAP. These results will impact the field because it departs markedly from the current inefficient, highly invasive method of physically removing surfactant by whole lung lavage (WLL) and instead uses a novel approach to restore AM function. This study is expected to establish the feasibility of a novel, specific therapy for children with hPAP and a new type of cell transplantation therapy (PMT) that may be useful for other diseases.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following conditions to be eligible for participation in this study:

1. Male or female with a confirmed diagnosis of hPAP defined as:

   * Homozygous or compound heterozygous CSF2RA mutations - AND -
   * A normal GM-CSF autoantibody test result - AND -
   * An abnormal STAT5-PI test result - OR -
   * An abnormal GM-CSF 50% effective concentration (EC50) test result
2. Diffuse ground glass opacification of the lungs visualized on a chest computed tomogram (CT)
3. History of prior receipt of WLL therapy or moderate hPAP lung disease severity requiring therapy in the opinion of the Clinical Site Investigator and/or Sponsor
4. Able to undergo bone marrow collection by routine clinical aspiration
5. 18 years of age or older on the date the Informed consent form (ICF) is signed
6. Females who have been post-menopausal for >2 years or females of child-bearing potential after a confirmed menstrual period using a highly efficient method of contraception (as described in Section 11.4.2) for the period from 3 months prior to the first administration of gene-corrected macrophages until 12 months after the last administration of gene-corrected macrophages. Females of child-bearing potential must have a negative serum pregnancy test at Screening (Visit 1), at bone marrow collection (Visit 2), and immediately before each administration of gene-corrected macrophages (Visits 3, 5, 7), and must not be lactating.
7. Males of reproductive potential must agree to use condoms for the period from the 1st administration of gene-corrected macrophages until 12 months after the last dose of gene-corrected macrophages, have a partner who is not of child-bearing potential (i.e. men or females who have been post-menopausal for >2 years), or have a female partner who is using adequate contraception as described in Section 11.4.2.
8. Signed written informed consent form (ICF)

Exclusion Criteria:

Patients who meet any of the following conditions will not be eligible for participation in this study:

1. History of a confirmed diagnosis of any other PAP-causing disease defined as:

   1. PAP caused by function-altering mutations in CSF2RB, adenosine triphosphate (ATP)-binding cassette subfamily A member 3 (ABCA3), SFTPB, SFTPC, Thyroid Transcription Factor 1 (TTF-1), GATA-binding factor 2 (GATA2), SLC7A7, and methionyl-transfer RNA (tRNA) synthetase (MARS), or other genes demonstrated to cause PAP other than CSF2RA
   2. PAP associated with an abnormal GM-CSF autoantibody test
   3. PAP associated with hematologic disorders including but not limited to myelodysplasia, aplastic anemia, leukemia, multiple myeloma, lymphoma
   4. PAP associated with non-hematologic malignancies
   5. PAP associated with immune deficiency syndromes
   6. PAP associated with chronic inflammatory syndromes
   7. PAP associated with chronic infections including but not limited to human immunodeficiency virus, Mycobacteria tuberculosis or other Mycobacterial species, or other organisms
   8. PAP associated with inhaled materials including but not limited to inorganic dusts (e.g., silica, titanium, indium, aluminum), organic dusts (e.g., sawdust, fertilizer); or gases/vapors (e.g., cleaning products, paints, and welding-related fumes)
2. Pulmonary fibrosis that is clinically significant in the opinion of Clinical Site Investigator and/or Sponsor
3. A confirmed (i.e., repeated) positive serum anti-GM-CSF receptor antibody test and/or a confirmed positive anti-lentiviral antibody test at the time of screening and prior to each administration of gene-corrected macrophages
4. History of receipt of any investigational agent within 3 months of Study Visit 3
5. History of active chronic infection (e.g., HIV, Hepatitis, others) at the time of Screening
6. History of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to Study Visit 3, defined as more than 14 drinks/week for females or 21 drinks/week for males (1 drink - 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer, or 1.5 ounces (45 ml) of hard liquor)
7. History of medication or illicit drug abuse within 1 year prior to Study Visit 3, including but not limited to cocaine, heroin, or other opioids
8. Currently or planning to become pregnant between the Screening visit and Visit 14 and/or currently breast-feeding
9. Any other medical, behavioral, or psychiatric condition that would interfere with the completion of Study Visits or assessments in the opinion of the Clinical Site Investigator and/or Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2038-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) | Pre- and Post-PMT Therapy for 15 years
  Number of patients with a CTCAE grade 3 or 4 AE in clinical history findings, physical exam findings, vital signs, clinical laboratory values, pulmonary function data, cardiac function, chest x-ray, chest CT at any time during the study period after initiation of PMT Therapy

SECONDARY OUTCOMES:
Tolerability of Pulmonary Macrophage Transplantation (PMT) Therapy | For 2 days prior to PMT, immediately upon completion of PMT, and daily for 5 days following each PMT procedure.
  Patient global impression of severity (PGIS) and patient global impression of change (PGIC) will be assessed in relation to the patient's overall impression of disease severity and change from baseline. PGIS will assess the current breathing problems and the impact on daily physical activity. The current severity of hPAP (PGIS) will be assessed on a five-point scale ranging from none, mild, moderate, severe, to very severe.
  PGIC will assess the change from baseline in breathing problems and impact of breathing problems on daily physical activity. The change from baseline in hPAP severity (PGIC) will be assessed on a five-point scale ranging from much improved, somewhat improved, no change, somewhat worse, to much worse.
  The PGIS and PGIC parameters will be evaluated just prior to PMT, immediately upon completion of PMT, and daily for 5 days following PMT.
Number of patients with an increase in anti-GM-CSF receptor alpha antibodies | Pre- and Post-PMT Therapy for 15 years
  Number of patients with an increase in detection of anti-GM-CSF receptor alpha antibodies in serum at any time during the study period after initiation of PMT Therapy
Number of patients with evidence of clonal lentiviral positive cell expansion | Pre- and Post-PMT Therapy for 15 years
  Number of patients with evidence of clonal lentiviral positive cell expansion measured by the presence of vector-derived replication competent lentivirus (RCL) at any time during the study period after initiation of PMT Therapy
Number of patients with lentiviral vector insertion site analysis indicative of clonal dominance or leukemia | Pre- and Post-PMT Therapy for 15 years
  Number of patients with evidence of insertion of the transgene in proximity of known proto-oncogenes and the number of patients with evidence of clonal expansion associated to common insertion sites at any time during the study period after initiation of PMT Therapy
Number of patients with increased biomarkers of inflammation in bronchoalveolar lavage (BAL) fluid or serum | Pre- and Post-PMT Therapy for 15 years
  Number of patients with a CTCAE grade 3 or 4 increase in tumor necrosis factor (TNF)-alpha, interleukin (IL)-1-beta, and IL-6 in bronchoalveolar lavage (BAL) or serum at any time during the study period after initiation of PMT Therapy
Percent of BAL cells with detectable GM-CSF Receptor Alpha Chain Expression | 16 months
  Change in the percentage of BAL cells with detectable GM-CSF receptor alpha chain expression measured by immunofluorescence at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Percent of proliferating alveolar macrophages | 16 months
  Change in percentage of alveolar macrophages that stain positive for Ki-67 at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Biodistribution of transplanted macrophages via detection of lentiviral DNA in BAL and blood | 16 months
  Presence of lentiviral DNA detected by PCR in the lungs and blood at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Durability of the Therapy - percent of GM-CSF Receptor Alpha Chain expressing alveolar macrophages | 6 months (Visit 11) and 12 months (Visit 14) after PMT Therapy
  Change in the percentage of BAL cells with detectable GM-CSF receptor alpha chain expression measured by immunofluorescence at 6 months (Visit 11) compared to one year after PMT Therapy (Visit 14)
Turbidity of the bronchoalveolar lavage fluid | 16 months
  Change in bronchoalveolar lavage (BAL) fluid turbidity at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Ratio of surfactant cholesterol to total phospholipid | 16 months
  Change in ratio of cholesterol to total phospholipids in surfactant at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Percentage of alveolar macrophages with neutral lipid accumulation | 16 months
  Change in the percentage of Oil Red O+ alveolar macrophages at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Intensity of AMs neutral lipid accumulation | 16 months
  Change in intensity of Oil Red O staining in AM at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16). Intensity will be graded on visual scoring. Each cell will be assigned a number (0, 1, 2, or 3) reflecting the degree of oil-red-O-staining. The number of cells at each grade will be multiplied by the numerical grade and products added and divided by the total number of cells evaluated to obtain the oil-red-O staining score.
Concentration of PAP biomarkers in bronchoalveolar lavage fluid | 16 months
  Change in concentrations of BAL cytokine biomarkers of PAP (GM-CSF, M-CSF, and monocyte chemotactic protein-1 (MCP-1)) measured by enzyme linked immunosorbent assay (ELISA) at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Difference in expression of alveolar macrophage mRNA biomarkers of Pulmonary Alveolar Proteinosis | 16 months
  Change in alveolar macrophage messenger RNA (mRNA) biomarkers of PAP (PU.1, peroxisome proliferator-activated receptor (PPAR)-gamma, and ABCG1) measured by quantitative reverse transcription/polymerase chain reaction (qRT-PCR) amplification at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Difference in alveolar-arterial difference in oxygen concentration (A-aDO2) | 16 months
  Change in A-aDO2 measured by standardized arterial blood gas analysis at baseline and at 6 months and one year after PMT Therapy
Difference in San Diego Shortness of Breath Questionnaire Score | 16 months
  Change in dyspnea measured by the San Diego Dyspnea Questionnaire at baseline and all visits after PMT
  The San Diego Dyspnea Questionnaire asks subjects to indicate severity of shortness of breath on a 6-point scale (0=Not at all, 5=maximally or unable to do because of breathlessness) during 21 activities of daily living associated with varying levels of exertion. Three additional questions ask about fear of harm from overexertion, limitations, and fear caused by shortness of breath, for a total of 24 items. A total sum score ranges from 0 to 120.
Difference in pulmonary oxygen delivery | 16 months
  Change in the diffusing capacity for carbon monoxide (DLCO) measured by American Thoracic Society (ATS) standards at baseline and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Difference in exercise-induced peripheral blood oxygen desaturation trough via treadmill test | 16 months
  Change in lowest peripheral blood oxygen saturation value measured by standardized treadmill testing performed at baseline and at 6 months and one year after PMT Therapy
Difference in time to exercise-induced peripheral blood oxygen desaturation via treadmill test | 16 months
  Change in time to reduction in peripheral blood oxygen saturation by 5% measured by standardized treadmill testing performed at baseline and at 6 months and one year after PMT Therapy
Difference in exercise-induced peripheral blood oxygen desaturation trough via STEP test | 16 months
  Change in lowest peripheral blood oxygen saturation value measured by the STandardized Exercise Protocol testing (STEP Test) performed weekly before and after initiation of PMT Therapy.
  Standardized exercise oximetry to measure blood oxygen saturation will be performed at home weekly during the study. Briefly, a pulse-oximeter will be placed on the finger with the participant at rest sitting in a chair. Three baseline (resting) readings will be taken over a 3 minute period. Then the participant will step on and off a standard step for a period of 5 minutes followed by a 3 minute seated recovery. The pulse oximeter will record oxygen saturations every minute of the test. Data will be transmitted to the site via the mobile health platform. The lowest peripheral blood oxygen saturation will be determined from the collected data.
Difference in time to exercise-induced peripheral blood oxygen desaturation via STEP test | 16 months
  Change in time to reduction in peripheral blood oxygen saturation (SpO2) by 5% measured by the STandardized Exercise Protocol testing (STEP Test) performed weekly before and after initiation of PMT Therapy. Results will be evaluated by repeated measures analysis and graphic illustration to depict temporal change in the therapeutic effects after PMT.
  Standardized exercise oximetry to measure blood oxygen saturation will be performed at home weekly during the study. Briefly, a pulse-oximeter will be placed on the finger with the participant at rest sitting in a chair. Three baseline (resting) readings will be taken over a 3-minute period. Then the participant will step on and off a standard step for a period of 5 minutes followed by a 3-minute seated recovery. The pulse oximeter will record oxygen saturations every minute of the test. Data will be transmitted to the site via the mobile health platform. The time of the lowest SpO2 will be determined from the collected data.
Difference in severity of lung disease via lung density via quantitative CT densitometry | 16 months
  Change in lung mass determined radiologically by quantitative pulmonary computed tomographic densitometry (QPCTD) at baseline and at 6 months and one year after PMT Therapy
Difference in severity of lung disease via pulmonary parenchymal pattern score | 16 months
  Change in the quantitative categorical pulmonary parenchymal pattern score determined using CALIPER at baseline and at 6 months and one year after PMT Therapy
Difference in Health Status/Quality of Life Score via the 36-Item Short Form Survey (SF-36) Questionnaire | 16 months
  Change in quality of life measured by SF-36 total score and component score at baseline (Visit 3) and all visits after PMT.
  The SF-36 Questionnaire is a 36-item, patient-reported survey of patient health. The questionnaire consists of eight scaled scores (each 0-100), which are the weighted sums of the questions in their section, with each question carrying equal weight. The lower the score the more disability. The eight sections are 1) vitality, 2) physical functioning, 3) bodily pain, 4) general health perceptions, 5) physical role functioning, 6) emotional role functioning, 7) social role functioning and 8) mental health.

OTHER OUTCOMES:
Percentage of bronchoalveolar lavage cells that respond to GM-CSF stimulation | 16 months
  Change in the percentage of BAL cells positive for phosphorylated STAT5 (pSTAT5) and change in STAT5 phosphorylation index (STAT5-PI) via flow cytometry at baseline (Visit 3) and various times after PMT (months 2, 4, 6 (optional), 10, and 16)
Cell population dynamics of transplanted macrophages via RNA sequencing t-distributed stochastic neighborhood embedding analysis (t-SNE) | 16 months
  Change in cell population dynamics of the transplanted macrophages following PMT Therapy using t-distributed stochastic neighbor embedding (t-SNE) analysis of RNA sequencing data obtained at single-cell resolution on cells collected by BAL (months 2, 4, 6 (optional), 10, and 16). Specifically, the investigators will track the number and relative proportion of distinct cell populations among BAL cells.
Transcriptional regulation of alveolar macrophage specification via an assay for transposable-accessible chromatin with sequencing | 16 months
  The upstream regulatory elements controlling downstream target genes regulating AM specification will be identified in transplanted macrophages collected by BAL (months 2, 4, 6 (optional), 10, and 16). Monocle and Cicero software will utilize a battery of regression analysis tools to identify and correlate differentially expressed genes and differentially accessible putative DNA regulatory elements.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Towe, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No